CLINICAL TRIAL: NCT00122694
Title: Modification of Chronic Inflammation by Inhaled Carbon Monoxide in Patients With Stable COPD
Brief Title: Modification of Chronic Inflammation by Inhaled Carbon Monoxide in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Collaborators: Stichting Astma Bestrijding, The Netherlands (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: METc2003.249; SAB 2004/024
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: carbon monoxide; COPD; inflammation; sputum induction; stable COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Carbon Monoxide

INTERVENTIONS:
Drug: carbon monoxide

SUMMARY:
The purpose of this study is to determine whether carbon monoxide is effective in the treatment of stable COPD.

DETAILED DESCRIPTION:
COPD is characterised by a chronic pulmonary inflammation and a shifted oxidant/antioxidant balance. The main cause of this inflammation is smoking. After smoking cessation, this inflammation and shifted oxidant/antioxidant balance continues. This causes an increased deterioration of lung function compared to healthy persons of matching age.

The ongoing inflammation appears to be relatively insensitive to corticosteroid therapy.

Until now, there is no therapy for this inflammation. Both in vitro and in vivo studies show that carbon monoxide has, besides an antioxidant capacity, anti-inflammatory properties. The aim of this trial is to study whether the inflammation can be reduced by inhalation of carbon monoxide.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age > 40 years. Women must be post-menopausal (i.e. at least one year must have passed after the last menstruation), surgically sterile or using acceptable contraceptives, as judged by the investigator.
* A diagnosis of COPD according to the criteria of the American Thoracic Society (ATS); a disease state characterised by the presence of chronic airway obstruction due to chronic bronchitis (cough/sputum on most days a week for 3 months a year for at least two successive years); or emphysema.
* FEV1 > 0.7 litres
* FEV1/FVC ratio < 70% (equation retrieval system [ERS] equations)
* A smoking history of > 10 pack years
* Completely stopped smoking > 1 year ago
* No upper or lower respiratory tract infection in the last 4 weeks
* In a stable phase of COPD, as judged by the investigator
* Signed and dated informed consent obtained before any study related procedures (including withdrawal of concomitant medication) are conducted

Exclusion Criteria:

* Treatment with immune-modulating agents for any other disease
* History of asthma; former diagnosis of asthma
* Arterial oxygen tension (PaO2) < 8.0 kPa
* Any significant other pulmonary disease or disorder (e.g. alpha1-antitrypsin deficiency, bronchiectasies), as judged by the investigator
* Patients with other significant disease or disorder (like cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic [including diagnosed diabetes], malignant, psychiatric, major physical impairment), which, in the opinion of the investigator may either put the patient at risk because of participation in the study; or may influence the results of the study, or the patient's ability to participate in the study.
* Patients unable to blow reproducable lung function measurements
* Patients using medicine with anti-oxidant character like n-acetyl-cysteine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-01; Study Completion 2006-03

PRIMARY OUTCOMES:
percentage of neutrophils in induced sputum

SECONDARY OUTCOMES:
methacholine provocation threshold
exhaled CO/NO
FEV1, FVC, RAW, sgaw
inflammatory parameters in sputum and blood
8-isoprostane in exhaled breath

CONTACTS AND LOCATIONS:
Overall Officials: H AM Kerstjens, Prof., MD, PhD, Principal Investigator — University Medical Center Groningen, Department of Pulmonary Diseases
Locations (1):
- University Medical Center Groningen, Department of Pulmonary Diseases, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Bathoorn E, Slebos DJ, Postma DS, Koeter GH, van Oosterhout AJ, van der Toorn M, Boezen HM, Kerstjens HA. Anti-inflammatory effects of inhaled carbon monoxide in patients with COPD: a pilot study. Eur Respir J. 2007 Dec;30(6):1131-7. doi: 10.1183/09031936.00163206. Epub 2007 Aug 22. PMID 17715164